CLINICAL TRIAL: NCT07292844
Title: Effect of Geranium Inhalation Aromatherapy on Reducing Pain and Blood Pressure Among Indonesian Cancer Patients Undergoing Chemotherapy: A Randomized Controlled Trial
Brief Title: Effect of Geranium Inhalation Aromatherapy on Pain and Blood Pressure in Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Surakarta (Other)
Responsible Party: Principal Investigator, Fahrun Nur Rosyid, Head of Quality Assurance Group, Universitas Muhammadiyah Surakarta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMS-GERANIUM-RCT2022
Record Dates: First submitted 2025-11-22; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Chemotherapy Induced Pain; Blood Pressure Changes in Cancer Patients; Chemotherapy Side Effects
Keywords: Blood Pressure; Cancer; Chemotherapy; Geranium Aromatherapy; Pain
MeSH Terms: conditions — Neoplasms; Pain | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into two parallel groups (geranium aromatherapy vs. control) with no crossover during the study period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geranium Inhalation Aromatherapy (Experimental): Participants in this arm received geranium inhalation aromatherapy during their chemotherapy session. Three drops of geranium essential oil were placed on a piece of cotton and inhaled for 15 minutes during chemotherapy, administered twice per month. Pain and blood pressure were assessed before and after the intervention
  Interventions: Other: Geranium Inhalation Aromatherapy
- Usual Care / No Aromatherapy (No Intervention): Participants in this arm received standard chemotherapy care without any aromatherapy intervention. They underwent the same assessment procedures as the intervention group, including pre- and post-treatment measurements of pain and blood pressure, but no essential oil was administered

INTERVENTIONS:
Other: Geranium Inhalation Aromatherapy — Participants received inhalation aromatherapy using geranium essential oil during their chemotherapy session. Three drops of geranium essential oil were placed on a piece of cotton positioned near the patient to allow continuous inhalation. The aromatherapy was administered for 15 minutes during chemotherapy and given twice per month. Pain intensity (VAS) and blood pressure were measured before and after each session. The control group received usual care without aromatherapy.
  Other Names: Geranium Essential Oil Inhalation; Aromatherapy with Geranium Oil
  Arms: Geranium Inhalation Aromatherapy

SUMMARY:
This randomized controlled trial aims to examine the effect of geranium inhalation aromatherapy on pain and blood pressure among Indonesian cancer patients undergoing intravenous chemotherapy. A total of 90 participants under the age of 65 with normal BMI will be enrolled and randomly assigned to either an intervention group or a control group. The intervention group will receive geranium essential oil inhalation using three drops applied to cotton and inhaled for 15 minutes during chemotherapy sessions, while the control group will receive usual care without aromatherapy. Pain intensity will be measured using the Visual Analog Scale (VAS), and blood pressure will be recorded using a standard digital blood pressure monitor before and after the intervention. This study aims to evaluate whether geranium aromatherapy can be feasibly implemented as a complementary supportive therapy during chemotherapy. Study Started Date after January 18, 2017

DETAILED DESCRIPTION:
Cancer patients undergoing chemotherapy frequently experience a range of physical and psychological side effects, including pain, fatigue, nausea, sleep disturbances, and fluctuations in blood pressure. Complementary approaches such as aromatherapy are increasingly explored as supportive interventions due to their accessibility, safety, and low cost. Geranium essential oil contains bioactive components such as geraniol and citronellol, which have been noted for potential analgesic, anti-inflammatory, and relaxing properties. This study utilizes a randomized controlled trial design to evaluate the effect of geranium inhalation aromatherapy on pain and blood pressure among cancer patients undergoing chemotherapy at a public hospital in Surakarta, Indonesia. Ethical approval was obtained from the Health Research Ethics Committee of Dr. Moewardi General Hospital prior to participant recruitment.

Ninety patients meeting the inclusion criteria (age < 65 years, normal BMI, undergoing chemotherapy regimen 1, and providing informed consent) will be selected using simple random sampling. Participants will be randomly assigned into two equal groups: an intervention group receiving geranium inhalation aromatherapy and a control group receiving standard care without aromatherapy. The intervention consists of applying three drops of geranium essential oil onto cotton, which patients will inhale for 15 minutes during their chemotherapy sessions, conducted twice per month. Pre- and post-intervention assessments will include demographic characteristics, pain intensity measured using the Visual Analog Scale (VAS), and blood pressure recorded using an OMRON digital blood pressure monitor. Data analysis will involve paired t-tests, independent t-tests, and chi-square tests, with statistical significance set at p < 0.05. This study is designed to explore potential physiological mechanisms related to aromatherapy, which may include olfactory system stimulation, relaxation responses, modulation of endogenous hormones, and autonomic regulation. The study also acknowledges possible limitations such as sample size, intervention duration, and the absence of biomarker assessments.

ELIGIBILITY:
Inclusion:

1. Cancer patients undergoing intravenous chemotherapy (regimen 1 / series 1)
2. Age less than 65 years
3. Body Mass Index (BMI) between 18.5 and 22.9 kg/m².
4. Willing to participate and able to provide informed consent.

Exlusion:

1. Patients with conditions affecting the sense of smell (e.g., severe nasal obstruction or anosmia).
2. Patients with known allergies to essential oils or plant-based aromatherapy products.
3. Patients experiencing acute medical emergencies or unstable hemodynamic conditions during chemotherapy.
4. Patients who withdraw consent at any stage of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity (Visual Analog Scale - VAS) | Measured immediately before and after each aromatherapy session (single-session pre-post measurement).
  Pain intensity was measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain). Measurements were conducted immediately before the intervention and immediately after the 15-minute aromatherapy exposure during chemotherapy. The primary outcome is the change in VAS score from pre- to post-intervention.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure | Measured immediately before and after each aromatherapy session.
  Diastolic blood pressure was measured using the OMRON HEM-7156AT blood pressure device before and after the 15-minute aromatherapy exposure. The outcome is defined as the pre-post change in diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: FIK UMS, Principal Investigator — Universitas Muhammadiyah Surakarta
Locations (1):
- RSUD Dr. Moewardi Surakarta, Surakarta, Centre Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study did not include a data sharing plan in the ethics approval, and the dataset contains identifiable clinical information that cannot be disclosed